CLINICAL TRIAL: NCT07146139
Title: MyPrEP Plus: Development and Pilot Testing of Novel Preexposure Prophylaxis Decision Support Tools for Transgender Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was halted prematurely as a result of the termination of the grant by the NIH.
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00083027
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HIV Pre-exposure Prophylaxis; HIV Prevention and Care; Mobile Health Technology (mHealth); Adherence; Doxycycline STI PEP
Keywords: PrEP; Pre-exposure prophylaxis; MyPrEP; Website; Decision Support
MeSH Terms: interventions — Drug Packaging; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with two participants randomized to the main study intervention (MyPrEP Plus) for every one participant randomized to PrEP support with the standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Conditon: MyPrEP Plus (Experimental): The intervention administered in the experimental condition includes PrEP decisional and adherence support with the MyPrEP Plus package.
  Interventions: Device: MyPrEP Plus Package
- Control Condition: Standard of Care (Other): Participants randomized to the control condition will receive PrEP support through the standard of care.
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Device: MyPrEP Plus Package — Participants receiving the MyPrEP Plus Package will utilize the interactive MyPrEP website to learn about PrEP and the various kinds of PrEP available as well as information about Doxy-PEP. While on PrEP, participants will be able sign up for PrEPmate, a tool designed to support PrEP adherence.
  Arms: Experimental Conditon: MyPrEP Plus
Behavioral: Standard of Care (SOC) — Participants in the control condition will receive PrEP support according to local standard of care while using the website pleaseprepme.org.
  Arms: Control Condition: Standard of Care

SUMMARY:
The primary goal of this randomized controlled trial is to learn if a decision support tool called MyPrEP Plus can help transgender women make decisions about taking pre-exposure prophylaxis (PrEP) for HIV prevention.

DETAILED DESCRIPTION:
In this clinical study, 60 transgender women will be randomly assigned to one of two groups, either PrEP support via standard of care through pleaseprepme.org (control condition) or PrEP support with the MyPrEP Plus package (experimental condition) which includes access to the MyPrEP website which provides information on the various types of PrEP as well as information on Doxy-PEP. Participants will also have access to PrEPmate, a two-way PrEP support tool that is meant to help participants stay engaged in their PrEP care and is meant to support starting PrEP and staying on PrEP.

Participants in each group will start out by completing a baseline questionnaire that will ask about demographics, behaviors, and PrEP and Doxy-PEP knowledge. Each participant will be followed for three months while deciding to take PrEP or actively taking PrEP. At the end of three months, participants will be administered another survey which will assess PrEP uptake, change in PrEP and Doxy-PEP knowledge, and how well the MyPrEP Plus package helped with starting and staying on PrEP. Around 20 participants in the experimental condition will be invited for an in-depth interview to discuss their experience using the MyPrEP Plus package.

ELIGIBILITY:
Inclusion Criteria:

* Are age 18 or older
* Identify as a transgender woman or woman and was assigned male sex at birth
* Are not currently on PrEP in the last three months and interested in learning more about PrEP
* Able to successfully send and receive text messages
* HIV negative by self-report
* Are able to speak, read and write in English or Spanish
* Report any of the following in the last 12 months:

  * Having anal or vaginal sex with a person assigned male at birth
  * Exchange of sex for money, goods, or services
  * Received a diagnosis of a sexually transmitted infection
  * Sharing injection equipment
* Are able and willing to provide written informed consent and participate for the duration of the study

Exclusion Criteria:

* In a mutually monogamous sexual relationship with an HIV-negative partner for the past 12 months
* Of any medical, psychiatric, or social condition that in the opinion of the investigator would preclude participation or their ability to remain in the trial
* Study site staff member

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender woman or woman and was assigned male sex at birth
Enrollment: 2 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the MyPrEP Plus package for PrEP uptake in TGW as assessed by the Client Satisfaction Questionnaire, System Usability Scale, and intervention metrics. | 3 months
  Participant responses to the Client Satisfaction Questionnaire (CSQ-8) and the System Usability Scale (SUS) assessment tools which assess the various domains of the combined tools will be used to evaluate the acceptability of the MyPrEP Plus package. Scores for the CSQ-8 and the SUS range from 8-32 and 0-100, respectively with higher scores representing greater satisfaction and usability. Web-based analytics of the MyPrEP website combined with responses within the PrEPmate tool and time spent using PrEPmate to interact with staff will be used as a measure of feasibility.

SECONDARY OUTCOMES:
Participants' change in knowledge of PrEP and doxycycline PEP (Doxy-PEP) after three months of study participation as assessed by a set of knowledge questions at baseline and follow up. | 3 months
  Participant responses to a series of true/false questions about PrEP and Doxy-PEP. Items assess knowledge of the various kinds of PrEP, knowledge of Doxy-PEP, how each type of PrEP is taken, conditions that Doxy-PEP can help prevent and common side effects of the various forms of PrEP as well as Doxy-PEP. Responses will be labeled as correct or incorrect. The change in the proportion of correct answers to the PrEP and Doxy-PEP knowledge questionnaire at three months from baseline will be calculated for each participant.
Preliminary impact of the MyPrEP Plus package on PrEP uptake in TGW compared to that of pleaseprepme.org by evaluating the number of people who access PrEP after 3 months. | 3 months
  The number of participants using the MyPrEP Plus Package vs. the number of participants using pleaseprepme.org who demonstrate PrEP uptake by confirming PrEP acquisition with a physical bottle for oral PrEP or documented administration of injectable PrEP.
Preliminary impact of the MyPrEP Plus package on Doxy-PEP uptake by evaluating the number of people who access Doxy-PEP after 3 months. | 3 months
  The number of participants using the MyPrEP Plus Package vs. the number of participants using pleaseprepme.org who demonstrate Doxy-PEP uptake by confirming Doxy-PEP acquisition with a physical bottle.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Buchbinder, MD, Principal Investigator — Bridge HIV, San Francisco Department of Public Health
Locations (1):
- Bridge HIV, San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No